CLINICAL TRIAL: NCT04907201
Title: Electrophysiological Assessment of Cryoneurotomy in Spastic Lower Limbs.
Brief Title: H-reflex in Spastic Lower Limb Cryoneurotomy
Status: Active, not recruiting | Type: Observational
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Mahdis Hashemi, Research Assistant, Vancouver Island Health Authority
Other Study IDs: H20-02294
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Muscle Spasticity
Keywords: spasticity; Lower limb; H reflex; Cryoneurotomy; Range of motion
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: A group pf 30 patients with lower limb spasticity who are already candidate for cryoneurotomy will be invited to have an extra electrophysiological test for participation in this study. The test will be done for both limbs for a better comparison.
  Interventions: Procedure: Cryoneurotomy
- Healthy participants: A group of 30 healthy participants will be invited as a control group, and they will have a single session of electrodiagnostic test for their lower limb in dominant side.

INTERVENTIONS:
Procedure: Cryoneurotomy — Cryoneurotomy or application of a low temperature probe with guidance of ultrasound which is offered to the patients with lower limbs refractory spasticity as a part of their medical cares.
  Other Names: nerve cryoablation
  Groups: Patients

SUMMARY:
Spasticity is a common complication after many upper motor neurone disorders. Many surgical techniques have been introduced for patients with refractory spasticity though they are not without peri-operative risks. Cryoneurotomy is another procedure which is cheaper, faster and less invasive in comparison to other surgical interventions. While many studies support the use of cryoneurotomy for pain relief, there are not much studies on use of cryoneurotomy to manage spasticity. The purpose of this study to measure the effect of tibial nerve cryoneurotomy on electrophysiological and clinical spasticity measures in adult patients with spastic equinovarus or equinus foot, who will receive this procedure as a part of their treatment based on spasticity treatment available guidelines. The results will provide us valuable information like how long cryoneurotomy is effective, before regeneration happens.

DETAILED DESCRIPTION:
Different surgical techniques, including muscle and tendon lengthening and neurotomy/neurectomy (surgical sectioning of a peripheral nerve) are reserved for patients with refractory spasticity.

Cryoneurotomy which involves direct application of a low temperature probe to a nerve is another procedure, which is cheaper, faster and less invasive than surgical intervention, for the treatment of refractory spasticity. While many studies support using of cold temperature in pain relief (Ilfeld BM, 2017, Friedman, T. 2012), there are not much studies on use of cryoneurotomy to manage spasticity.This clinic has been using cryoneurotomy clinically with empiric success for 2.5 years. The initial results reveal significant increased active and passive range of motion in upper limbs and decreased clonus and improved gait after tibial neurotomy in lower limbs.

Spastic equinovarus foot (SEF) which is a common type of lower limb spasticity is typically treated with focal botulinum toxin injections, bracing and therapeutic exercise, although the drawback of these treatments is the need for serial injections and frequent interactions with health care providers. Recently selective tibial neurotomy has been shown to more definitively treat SEF (Bollens B, et al.2011, Deltombe T, et al. 2015), but as mentioned above this is an invasive approach. In light of our promising clinical experience with cryoneurotomy, we propose to prospectively and systematically measure its effect on SEF, as an alternative to more invasive surgical procedures and the typical multi-modal approach.

The data collection fro this project which is a single-centre, prospective cohort study will occur at the Victoria General Hospital (VGH) multidisciplinary spasticity clinic. Patients with spasticity are referred to this clinic for different procedures including cryoneurotomy. This study will not interfere or change the patients' medical care, and the assessments will be done for the patients who are already candidates for this procedure as a part of their treatment, besides other provided medical cares and have been accepted to receive that.These participants will be invited to have an extra electrophysiological test for being enrolled in this study, which will be performed before the procedure and at 1, 3 and 12 months after cryoneurotomy. In addition, the results of their routine physical examinations including spasticity degree and ankle passive range of motion will be collected in this study.

ELIGIBILITY:
Inclusion Criteria for patient group:

1. Patients who will have cryoneurotomy as part of their standard treatment for spastic equinovarus foot in VGH spasticity multidisciplinary clinic
2. Adults 18-70 years of age (male and female)
3. Ability to attend testing sessions, comply with testing protocols and provide written informed consent.
4. Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).

Inclusion Criteria for healthy participants:

1. Any healthy participants with the age between 18 to 70. Over 70 will be excluded due to the expected natural alterations in electrophysiological parameters
2. Able to attend and comply with the testing protocols
3. Able to provide informed written consent
4. Able to understand and speak English or have access to an appropriate interpreter

Exclusion Criteria:

1. History of previous nerve procedures such as chemical neurolysis with alcohol, cryoneurotomy, any surgery of the tibial nerve.
2. Any other neurological pathology different from that responsible for the spasticity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any adult patient with lower limb spasticity who is already candidate for cryoneurotmy as a part of their medical care will be asked to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Any changes in H max to M max amplitude ratio (H/ M ratio) | up to 12 months
  The ratio of maximum H reflex amplitude to maximum M wave amplitude as another electrophysiological analog for spasticity will be measured by a commercially available clinical electrodiagnosis machine before the procedure and at 1, 3 and 12 months after it. The results will be presented as a ratio and percentage.
Changes in maximum H reflex amplitude | up to 12 months after procedure
  The maximum H reflex amplitude as an analog of spasticity as it measure excitability of the monosynaptic reflex arc will be assessed by a commercially available clinical electrodiagnosis machine. The assessment will be done before the procedure and at 1, 3 and 12 months after it and at both sides. The measurement unit will be millivolt (mV).

SECONDARY OUTCOMES:
Degree of changes in ankle dorsi-flexion spasticity as measured by Modified Ashworth Scale (MAS) | up to 12 months after procedure
  MAS has 6 scales from 0 to 4 (0,1,1+,2,3,4) which 0 means no spasticity and 4 means the maximum spasticity and the affected limb is rigid in its position.The assessment will be done by a trained examiner which is not enrolled in providing medical care and will be done before the procedure and at 1, 3 and 12 months after the procedure.
Degree of changes in ankle dorsiflexion range of motion | Up to 12 months
  The active and maximum passive dorsiflexion range of motion will be measured by a goniometer and will be presented in degree. The test will be done before and at 1, 3 and 12 months after the procedure by a trained examiner who is not enrolled in providing medical care.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria General Hospital, Victoria, British Columbia, Canada

REFERENCES:
- [Background] Bollens B, Deltombe T, Detrembleur C, Gustin T, Stoquart G, Lejeune TM. Effects of selective tibial nerve neurotomy as a treatment for adults presenting with spastic equinovarus foot: a systematic review. J Rehabil Med. 2011 Mar;43(4):277-82. doi: 10.2340/16501977-0786. PMID 21305231
- [Background] Deltombe T, Bleyenheuft C, Gustin T. Comparison between tibial nerve block with anaesthetics and neurotomy in hemiplegic adults with spastic equinovarus foot. Ann Phys Rehabil Med. 2015 Apr;58(2):54-9. doi: 10.1016/j.rehab.2014.12.003. Epub 2015 Jan 9. PMID 25614022
- [Background] Friedman T, Richman D, Adler R. Sonographically guided cryoneurolysis: preliminary experience and clinical outcomes. J Ultrasound Med. 2012 Dec;31(12):2025-34. doi: 10.7863/jum.2012.31.12.2025. PMID 23197557
- [Background] Ilfeld BM, Gabriel RA, Trescot AM. Ultrasound-guided percutaneous cryoneurolysis for treatment of acute pain: could cryoanalgesia replace continuous peripheral nerve blocks? Br J Anaesth. 2017 Oct 1;119(4):703-706. doi: 10.1093/bja/aex142. No abstract available. PMID 29121277

DOCUMENTS (2):
  • Informed Consent Form: Control group (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04907201/ICF_000.pdf
  • Informed Consent Form: Patient group (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04907201/ICF_001.pdf